CLINICAL TRIAL: NCT02409680
Title: Aspirin Supplementation for Pregnancy Indicated Risk Reduction In Nulliparas (ASPIRIN)
Acronym: ASPIRIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Thomas Jefferson University (Other); Jawaharlal Nehru Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP ASPIRIN
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Results first posted 2021-09-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Premature Birth
Keywords: Preterm birth; Low dose aspirin
MeSH Terms: conditions — Premature Birth | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Active Comparator): Women will be randomized equally to receive daily low dose aspirin (LDA) [also known as acetylsalicylic acid (ASA)] of 81 mg beginning between 6 0/7 weeks and 13 6/7 weeks GA and continuing until 36 0/7 weeks GA or delivery.
  Interventions: Drug: Low dose aspirin
- Placebo Arm (Placebo Comparator): Women will be randomized equally to receive an identical appearing placebo beginning between 6 0/7 weeks and 13 6/7 weeks GA and continuing until 36 0/7 weeks GA or delivery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose aspirin — Daily administration of low dose (81 mg) aspirin [also known as acetylsalicylic acid (ASA], initiated between 6 0/7 weeks and 13 6/7 weeks GA and continued to 36 0/7 weeks GA compared to an identical appearing placebo. Compliance and outcomes will be assessed biweekly.
  Other Names: Acetylsalicylic acid (ASA)
  Arms: Intervention Arm
Drug: Placebo — Placebo
  Arms: Placebo Arm

SUMMARY:
Available data suggest that low dose aspirin may be a safe, widely available and inexpensive intervention that may significantly reduce the risk of preterm birth. However, this possibility needs to be proven in a properly designed randomized controlled trial (RCT) with preterm birth as the primary outcome. Such a clinical trial in a racially, ethnically and geographically diverse population could best be accomplished by the established infrastructure of the Global Network for Women's and Children's Health Research (GN).

DETAILED DESCRIPTION:
Background: Preterm birth (PTB) remains the leading cause of neonatal mortality and long term disability throughout the developed and developing world. Though complex in its origins, a growing body of evidence suggests that first trimester administration of low dose aspirin (LDA) holds promise to reduce the rate of PTB substantially.

Hypothesis: The investigators' primary hypothesis is that nulliparous women with no more than two previous first trimester pregnancy losses who are treated with LDA daily beginning between 6 0/7 weeks and 13 6/7 weeks gestational age (GA) through 36 0/7 weeks GA will reduce the risk of preterm birth from all causes.

Study Design Type: Prospective randomized, placebo-controlled, double-blinded multicenter clinical trial (patient level 1:1).

Population: Nulliparous women between the ages of 18 (or local age of majority) and 40 with no more than two previous first trimester pregnancy losses or any second trimester spontaneous pregnancy loss, a singleton pregnancy between 6 0/7 weeks and 13 6/7 weeks GA confirmed by ultrasound, and no contraindications to aspirin. Other medical conditions, such as sickle-cell anemia, may be considered a contraindication per the judgment of the site investigator.

Intervention: Daily administration of low dose (81 mg) aspirin [also known as acetylsalicylic acid (ASA)], initiated between 6 0/7 weeks and 13 6/7 weeks GA and continued to 36 0/7 weeks GA compared to an identical appearing placebo. Compliance and outcomes will be assessed biweekly.

Outcomes:

The primary outcome is to determine whether daily LDA initiated between 6 0/7 weeks and 13 6/7 weeks and continued to 36 0/7 weeks reduces the risk of preterm birth (birth prior to 37 0/7 weeks of pregnancy) by 20%. This will be determined based on assessed date of delivery in comparison to the projected estimated date of delivery, independent of whether or not the preterm delivery is indicated or spontaneous.

Secondary outcomes include:

* Preeclampsia and eclampsia (hypertensive disorders of pregnancy)
* Small for gestational age
* Perinatal mortality

Other secondary outcomes of interest are:

Maternal outcomes:

* Vaginal bleeding
* Antepartum hemorrhage
* Postpartum hemorrhage
* Maternal mortality
* Late abortion
* Change in maternal hemoglobin
* Preterm, preeclampsia

Fetal outcomes:

* Preterm birth <34 0/7 weeks of pregnancy
* Birth weight <2500g and <1500g
* Fetal loss
* Spontaneous abortion
* Stillbirth
* Medical termination of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women between 18 - 40 years of age. Minors who are ≥ 14 years of age may be enrolled if permitted by the country's ethical guidelines.
* No more than two previous first trimester pregnancy losses
* No medical contraindications to aspirin;
* Single live intrauterine pregnancy (IUP) between 6 0/7 and 13 6/7 weeks GA corroborated by an early dating ultrasound and with presence of a heartbeat.

Exclusion Criteria:

* Women prescribed daily aspirin for more than 7 days;
* Multiple gestations;
* Fetal anomaly by ultrasound (Note most fetal anomalies are not detectable by ultrasounds done at this early gestation. Subsequent discovery of a fetal anomaly is not viewed as an exclusion.);
* Hemoglobin < 7.0 gm/dl at screening;
* Any other medical conditions that may be considered a contraindication per the judgment of the site investigator (e.g., Lupus, Type 1 Diabetes, or any other known significant disease)
* Blood pressure ≥ 140/90 (Systolic blood pressure ≥ 140 and diastolic ≥ 90 at screening)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11976 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Koso-Thomas, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (14):
- United States (7):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of Colorado, Denver, Denver, Colorado
  - Indiana University, Indianapolis, Indiana
  - Boston University, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- Institute of Nutrition of Central America and Panama (INCAP), Guatemala City, Guatemala
- India (2):
  - KLE University's Jawaharlal Nehru Medical College, Belagavi, Karnataka
  - Lata Medical Research Foundation, Nagpur
- Moi University School of Medicine, Eldoret, Kenya
- The Aga Khan University, Karachi, Pakistan
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Background] Abramovici A, Cantu J, Jenkins SM. Tocolytic therapy for acute preterm labor. Obstet Gynecol Clin North Am. 2012 Mar;39(1):77-87. doi: 10.1016/j.ogc.2011.12.003. Epub 2012 Jan 4. PMID 22370109
- [Background] Ananth CV, Joseph KS, Oyelese Y, Demissie K, Vintzileos AM. Trends in preterm birth and perinatal mortality among singletons: United States, 1989 through 2000. Obstet Gynecol. 2005 May;105(5 Pt 1):1084-91. doi: 10.1097/01.AOG.0000158124.96300.c7. PMID 15863548
- [Background] Anderson RN, Smith BL. Deaths: leading causes for 2001. Natl Vital Stat Rep. 2003 Nov 7;52(9):1-85. PMID 14626726
- [Background] Baschat AA, Guclu S, Kush ML, Gembruch U, Weiner CP, Harman CR. Venous Doppler in the prediction of acid-base status of growth-restricted fetuses with elevated placental blood flow resistance. Am J Obstet Gynecol. 2004 Jul;191(1):277-84. doi: 10.1016/j.ajog.2003.11.028. PMID 15295379
- [Background] Beck S, Wojdyla D, Say L, Betran AP, Merialdi M, Requejo JH, Rubens C, Menon R, Van Look PF. The worldwide incidence of preterm birth: a systematic review of maternal mortality and morbidity. Bull World Health Organ. 2010 Jan;88(1):31-8. doi: 10.2471/BLT.08.062554. Epub 2009 Sep 25. PMID 20428351
- [Background] Becker DM, Segal J, Vaidya D, Yanek LR, Herrera-Galeano JE, Bray PF, Moy TF, Becker LC, Faraday N. Sex differences in platelet reactivity and response to low-dose aspirin therapy. JAMA. 2006 Mar 22;295(12):1420-7. doi: 10.1001/jama.295.12.1420. PMID 16551714
- [Background] Bower SJ, Harrington KF, Schuchter K, McGirr C, Campbell S. Prediction of pre-eclampsia by abnormal uterine Doppler ultrasound and modification by aspirin. Br J Obstet Gynaecol. 1996 Jul;103(7):625-9. doi: 10.1111/j.1471-0528.1996.tb09829.x. PMID 8688387
- [Background] CAST: randomised placebo-controlled trial of early aspirin use in 20,000 patients with acute ischaemic stroke. CAST (Chinese Acute Stroke Trial) Collaborative Group. Lancet. 1997 Jun 7;349(9066):1641-9. PMID 9186381
- [Background] Chavarria ME, Lara-Gonzalez L, Gonzalez-Gleason A, Garcia-Paleta Y, Vital-Reyes VS, Reyes A. Prostacyclin/thromboxane early changes in pregnancies that are complicated by preeclampsia. Am J Obstet Gynecol. 2003 Apr;188(4):986-92. doi: 10.1067/mob.2003.203. PMID 12712098
- [Background] Chien PF, Arnott N, Gordon A, Owen P, Khan KS. How useful is uterine artery Doppler flow velocimetry in the prediction of pre-eclampsia, intrauterine growth retardation and perinatal death? An overview. BJOG. 2000 Feb;107(2):196-208. doi: 10.1111/j.1471-0528.2000.tb11690.x. PMID 10688503
- [Background] CLASP: a randomised trial of low-dose aspirin for the prevention and treatment of pre-eclampsia among 9364 pregnant women. CLASP (Collaborative Low-dose Aspirin Study in Pregnancy) Collaborative Group. Lancet. 1994 Mar 12;343(8898):619-29. PMID 7906809
- [Background] ACOG committee opinion no. 561: Nonmedically indicated early-term deliveries. Obstet Gynecol. 2013 Apr;121(4):911-915. doi: 10.1097/01.AOG.0000428649.57622.a7. PMID 23635710
- [Background] Coomarasamy A, Braunholtz D, Song F, Taylor R, Khan KS. Individualising use of aspirin to prevent pre-eclampsia: a framework for clinical decision making. BJOG. 2003 Oct;110(10):882-8. No abstract available. PMID 14550356
- [Background] Coomarasamy A, Honest H, Papaioannou S, Gee H, Khan KS. Aspirin for prevention of preeclampsia in women with historical risk factors: a systematic review. Obstet Gynecol. 2003 Jun;101(6):1319-32. doi: 10.1016/s0029-7844(03)00169-8. PMID 12798543
- [Background] Duley L, Henderson-Smart DJ, Knight M, King JF. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2004;(1):CD004659. doi: 10.1002/14651858.CD004659. PMID 14974075
- [Background] Duley L, Henderson-Smart DJ, Meher S, King JF. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004659. doi: 10.1002/14651858.CD004659.pub2. PMID 17443552
- [Background] Ebrashy A, Ibrahim M, Marzook A, Yousef D. Usefulness of aspirin therapy in high-risk pregnant women with abnormal uterine artery Doppler ultrasound at 14-16 weeks pregnancy: randomized controlled clinical trial. Croat Med J. 2005 Oct;46(5):826-31. PMID 16158479
- [Background] Erkan D, Merrill JT, Yazici Y, Sammaritano L, Buyon JP, Lockshin MD. High thrombosis rate after fetal loss in antiphospholipid syndrome: effective prophylaxis with aspirin. Arthritis Rheum. 2001 Jun;44(6):1466-7. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-C. No abstract available. PMID 11407709
- [Background] FitzGerald GA, Oates JA, Hawiger J, Maas RL, Roberts LJ 2nd, Lawson JA, Brash AR. Endogenous biosynthesis of prostacyclin and thromboxane and platelet function during chronic administration of aspirin in man. J Clin Invest. 1983 Mar;71(3):676-88. doi: 10.1172/jci110814. PMID 6338043
- [Background] Goffinet F, Aboulker D, Paris-Llado J, Bucourt M, Uzan M, Papiernik E, Breart G. Screening with a uterine Doppler in low risk pregnant women followed by low dose aspirin in women with abnormal results: a multicenter randomised controlled trial. BJOG. 2001 May;108(5):510-8. doi: 10.1111/j.1471-0528.2001.00116.x. PMID 11368138
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Goldenberg RL, Rouse DJ. Prevention of premature birth. N Engl J Med. 1998 Jul 30;339(5):313-20. doi: 10.1056/NEJM199807303390506. No abstract available. PMID 9682045
- [Background] Hamilton BE, Martin JA, Ventura SJ. Births: preliminary data for 2012. Natl Vital Stat Rep. 2013 Sep;62(3):1-20. PMID 24321416
- [Background] Heyborne KD. Preeclampsia prevention: lessons from the low-dose aspirin therapy trials. Am J Obstet Gynecol. 2000 Sep;183(3):523-8. doi: 10.1067/mob.2000.106757. PMID 10992168
- [Background] Kajantie E, Eriksson JG, Osmond C, Thornburg K, Barker DJ. Pre-eclampsia is associated with increased risk of stroke in the adult offspring: the Helsinki birth cohort study. Stroke. 2009 Apr;40(4):1176-80. doi: 10.1161/STROKEAHA.108.538025. Epub 2009 Mar 5. PMID 19265049
- [Background] Kim YJ, Lee BE, Park HS, Kang JG, Kim JO, Ha EH. Risk factors for preterm birth in Korea: a multicenter prospective study. Gynecol Obstet Invest. 2005;60(4):206-12. doi: 10.1159/000087207. Epub 2005 Jul 26. PMID 16088197
- [Background] Knight M, Duley L, Henderson-Smart DJ, King JF. Antiplatelet agents for preventing and treating pre-eclampsia. Cochrane Database Syst Rev. 2000;(2):CD000492. doi: 10.1002/14651858.CD000492. PMID 10796208
- [Background] Kozer E, Nikfar S, Costei A, Boskovic R, Nulman I, Koren G. Aspirin consumption during the first trimester of pregnancy and congenital anomalies: a meta-analysis. Am J Obstet Gynecol. 2002 Dec;187(6):1623-30. doi: 10.1067/mob.2002.127376. PMID 12501074
- [Background] Landau D, Shelef I, Polacheck H, Marks K, Holcberg G. Perinatal vasoconstrictive renal insufficiency associated with maternal nimesulide use. Am J Perinatol. 1999;16(9):441-4. doi: 10.1055/s-1999-6810. PMID 10774758
- [Background] Landolfi R, Cipriani MC, Novarese L. Thrombosis and bleeding in polycythemia vera and essential thrombocythemia: pathogenetic mechanisms and prevention. Best Pract Res Clin Haematol. 2006;19(3):617-33. doi: 10.1016/j.beha.2005.07.011. PMID 16781491
- [Background] Li DK, Liu L, Odouli R. Exposure to non-steroidal anti-inflammatory drugs during pregnancy and risk of miscarriage: population based cohort study. BMJ. 2003 Aug 16;327(7411):368. doi: 10.1136/bmj.327.7411.368. PMID 12919986
- [Background] Loe SM, Sanchez-Ramos L, Kaunitz AM. Assessing the neonatal safety of indomethacin tocolysis: a systematic review with meta-analysis. Obstet Gynecol. 2005 Jul;106(1):173-9. doi: 10.1097/01.AOG.0000168622.56478.df. PMID 15994634
- [Background] Low-dose aspirin in prevention and treatment of intrauterine growth retardation and pregnancy-induced hypertension. Italian study of aspirin in pregnancy. Lancet. 1993 Feb 13;341(8842):396-400. PMID 8094168
- [Background] March of Dimes, Save the Children, WHO. (2012). Born Too Soon: The Global Action Report on Preterm Birth. (M. V. K. CP Howson JE Lawn., Ed.). Geneva: World Health Organization.
- [Background] Marret S, Marchand L, Kaminski M, Larroque B, Arnaud C, Truffert P, Thirez G, Fresson J, Roze JC, Ancel PY; EPIPAGE Study Group. Prenatal low-dose aspirin and neurobehavioral outcomes of children born very preterm. Pediatrics. 2010 Jan;125(1):e29-34. doi: 10.1542/peds.2009-0994. Epub 2009 Dec 21. PMID 20026499
- [Background] Mathews TJ, Menacker F, MacDorman MF; Centers for Disease Control and Prevention, National Center for Health Statistics. Infant mortality statistics from the 2002 period: linked birth/infant death data set. Natl Vital Stat Rep. 2004 Nov 24;53(10):1-29. PMID 15622996
- [Background] McCormick MC, Richardson DK. Premature infants grow up. N Engl J Med. 2002 Jan 17;346(3):197-8. doi: 10.1056/NEJM200201173460310. No abstract available. PMID 11796855
- [Background] Morris JM, Fay RA, Ellwood DA, Cook CM, Devonald KJ. A randomized controlled trial of aspirin in patients with abnormal uterine artery blood flow. Obstet Gynecol. 1996 Jan;87(1):74-8. doi: 10.1016/0029-7844(95)00340-1. PMID 8532271
- [Background] Newnham JP, Godfrey M, Walters BJ, Phillips J, Evans SF. Low dose aspirin for the treatment of fetal growth restriction: a randomized controlled trial. Aust N Z J Obstet Gynaecol. 1995 Nov;35(4):370-4. doi: 10.1111/j.1479-828x.1995.tb02144.x. PMID 8717556
- [Background] Norgard B, Puho E, Czeizel AE, Skriver MV, Sorensen HT. Aspirin use during early pregnancy and the risk of congenital abnormalities: a population-based case-control study. Am J Obstet Gynecol. 2005 Mar;192(3):922-3. doi: 10.1016/j.ajog.2004.10.598. PMID 15746692
- [Background] Norton ME, Merrill J, Cooper BA, Kuller JA, Clyman RI. Neonatal complications after the administration of indomethacin for preterm labor. N Engl J Med. 1993 Nov 25;329(22):1602-7. doi: 10.1056/NEJM199311253292202. PMID 8232428
- [Background] Papageorghiou AT, Yu CK, Erasmus IE, Cuckle HS, Nicolaides KH. Assessment of risk for the development of pre-eclampsia by maternal characteristics and uterine artery Doppler. BJOG. 2005 Jun;112(6):703-9. doi: 10.1111/j.1471-0528.2005.00519.x. PMID 15924523
- [Background] Patrono C, Garcia Rodriguez LA, Landolfi R, Baigent C. Low-dose aspirin for the prevention of atherothrombosis. N Engl J Med. 2005 Dec 1;353(22):2373-83. doi: 10.1056/NEJMra052717. No abstract available. PMID 16319386
- [Background] Peruzzi L, Gianoglio B, Porcellini MG, Coppo R. Neonatal end-stage renal failure associated with maternal ingestion of cyclo-oxygenase-type-1 selective inhibitor nimesulide as tocolytic. Lancet. 1999 Nov 6;354(9190):1615. doi: 10.1016/S0140-6736(99)03105-0. PMID 10560684
- [Background] Physicians' health study: aspirin and primary prevention of coronary heart disease. N Engl J Med. 1989 Dec 28;321(26):1825-8. doi: 10.1056/NEJM198912283212610. No abstract available. PMID 2594041
- [Background] RE, B., & AS, B. (2006). Preterm Birth: Causes, Consequences, and Prevention. (I. of M. of the Academies, Ed.). Washington, DC: The National Academies Press.
- [Background] Ridker PM, Cook NR, Lee IM, Gordon D, Gaziano JM, Manson JE, Hennekens CH, Buring JE. A randomized trial of low-dose aspirin in the primary prevention of cardiovascular disease in women. N Engl J Med. 2005 Mar 31;352(13):1293-304. doi: 10.1056/NEJMoa050613. Epub 2005 Mar 7. PMID 15753114
- [Background] Saigal S, Doyle LW. An overview of mortality and sequelae of preterm birth from infancy to adulthood. Lancet. 2008 Jan 19;371(9608):261-9. doi: 10.1016/S0140-6736(08)60136-1. PMID 18207020
- [Background] Schisterman EF, Silver RM, Lesher LL, Faraggi D, Wactawski-Wende J, Townsend JM, Lynch AM, Perkins NJ, Mumford SL, Galai N. Preconception low-dose aspirin and pregnancy outcomes: results from the EAGeR randomised trial. Lancet. 2014 Jul 5;384(9937):29-36. doi: 10.1016/S0140-6736(14)60157-4. Epub 2014 Apr 2. PMID 24702835
- [Background] Seamon LG, Cohn DE, Henretta MS, Kim KH, Carlson MJ, Phillips GS, Fowler JM. Minimally invasive comprehensive surgical staging for endometrial cancer: Robotics or laparoscopy? Gynecol Oncol. 2009 Apr;113(1):36-41. doi: 10.1016/j.ygyno.2008.12.005. Epub 2009 Jan 24. PMID 19168206
- [Background] Silver RM, Edwin SS, Trautman MS, Simmons DL, Branch DW, Dudley DJ, Mitchell MD. Bacterial lipopolysaccharide-mediated fetal death. Production of a newly recognized form of inducible cyclooxygenase (COX-2) in murine decidua in response to lipopolysaccharide. J Clin Invest. 1995 Feb;95(2):725-31. doi: 10.1172/JCI117719. PMID 7860753
- [Background] Smith GC. Life-table analysis of the risk of perinatal death at term and post term in singleton pregnancies. Am J Obstet Gynecol. 2001 Feb;184(3):489-96. doi: 10.1067/mob.2001.109735. PMID 11228508
- [Background] Smith GC, Shah I, Pell JP, Crossley JA, Dobbie R. Maternal obesity in early pregnancy and risk of spontaneous and elective preterm deliveries: a retrospective cohort study. Am J Public Health. 2007 Jan;97(1):157-62. doi: 10.2105/AJPH.2005.074294. Epub 2006 Nov 30. PMID 17138924
- [Background] Souter D, Harding J, McCowan L, O'Donnell C, McLeay E, Baxendale H. Antenatal indomethacin--adverse fetal effects confirmed. Aust N Z J Obstet Gynaecol. 1998 Feb;38(1):11-6. doi: 10.1111/j.1479-828x.1998.tb02949.x. PMID 9521382
- [Background] Subtil D, Goeusse P, Houfflin-Debarge V, Puech F, Lequien P, Breart G, Uzan S, Quandalle F, Delcourt YM, Malek YM; Essai Regional Aspirine Mere-Enfant (ERASME) Collaborative Group. Randomised comparison of uterine artery Doppler and aspirin (100 mg) with placebo in nulliparous women: the Essai Regional Aspirine Mere-Enfant study (Part 2). BJOG. 2003 May;110(5):485-91. doi: 10.1046/j.1471-0528.2003.t01-1-02097.x. PMID 12742333
- [Background] Vainio M, Kujansuu E, Iso-Mustajarvi M, Maenpaa J. Low dose acetylsalicylic acid in prevention of pregnancy-induced hypertension and intrauterine growth retardation in women with bilateral uterine artery notches. BJOG. 2002 Feb;109(2):161-7. doi: 10.1111/j.1471-0528.2002.01046.x. PMID 11888098
- [Background] Vainio M, Riutta A, Koivisto AM, Maenpaa J. Prostacyclin, thromboxane A and the effect of low-dose ASA in pregnancies at high risk for hypertensive disorders. Acta Obstet Gynecol Scand. 2004 Dec;83(12):1119-23. doi: 10.1111/j.0001-6349.2004.00396.x. PMID 15548142
- [Background] Valero De Bernabe J, Soriano T, Albaladejo R, Juarranz M, Calle ME, Martinez D, Dominguez-Rojas V. Risk factors for low birth weight: a review. Eur J Obstet Gynecol Reprod Biol. 2004 Sep 10;116(1):3-15. doi: 10.1016/j.ejogrb.2004.03.007. PMID 15294360
- [Background] Van Marter LJ, Leviton A, Allred EN, Pagano M, Sullivan KF, Cohen A, Epstein MF. Persistent pulmonary hypertension of the newborn and smoking and aspirin and nonsteroidal antiinflammatory drug consumption during pregnancy. Pediatrics. 1996 May;97(5):658-63. PMID 8628603
- [Background] Vane JR, Botting RM. The mechanism of action of aspirin. Thromb Res. 2003 Jun 15;110(5-6):255-8. doi: 10.1016/s0049-3848(03)00379-7. PMID 14592543
- [Background] Vermillion ST, Robinson CJ. Antiprostaglandin drugs. Obstet Gynecol Clin North Am. 2005 Sep;32(3):501-17. doi: 10.1016/j.ogc.2005.04.006. PMID 16125046
- [Background] Werler MM, Sheehan JE, Mitchell AA. Maternal medication use and risks of gastroschisis and small intestinal atresia. Am J Epidemiol. 2002 Jan 1;155(1):26-31. doi: 10.1093/aje/155.1.26. PMID 11772781
- [Background] Yu Y, Cheng Y, Fan J, Chen XS, Klein-Szanto A, Fitzgerald GA, Funk CD. Differential impact of prostaglandin H synthase 1 knockdown on platelets and parturition. J Clin Invest. 2005 Apr;115(4):986-95. doi: 10.1172/JCI23683. Epub 2005 Mar 17. PMID 15776109
- [Derived] Bucher S, Nowak K, Otieno K, Tenge C, Marete I, Rutto F, Kemboi M, Achieng E, Ekhaguere OA, Nyongesa P, Esamai FO, Liechty EA. Birth weight and gestational age distributions in a rural Kenyan population. BMC Pediatr. 2023 Mar 8;23(1):112. doi: 10.1186/s12887-023-03925-2. PMID 36890485
- [Derived] Hoffman MK, Goudar SS, Kodkany BS, Metgud M, Somannavar M, Okitawutshu J, Lokangaka A, Tshefu A, Bose CL, Mwapule A, Mwenechanya M, Chomba E, Carlo WA, Chicuy J, Figueroa L, Garces A, Krebs NF, Jessani S, Zehra F, Saleem S, Goldenberg RL, Kurhe K, Das P, Patel A, Hibberd PL, Achieng E, Nyongesa P, Esamai F, Liechty EA, Goco N, Hemingway-Foday J, Moore J, Nolen TL, McClure EM, Koso-Thomas M, Miodovnik M, Silver R, Derman RJ; ASPIRIN Study Group. Low-dose aspirin for the prevention of preterm delivery in nulliparous women with a singleton pregnancy (ASPIRIN): a randomised, double-blind, placebo-controlled trial. Lancet. 2020 Jan 25;395(10220):285-293. doi: 10.1016/S0140-6736(19)32973-3. PMID 31982074
- [Derived] Hoffman MK, Goudar SS, Kodkany BS, Goco N, Koso-Thomas M, Miodovnik M, McClure EM, Wallace DD, Hemingway-Foday JJ, Tshefu A, Lokangaka A, Bose CL, Chomba E, Mwenechanya M, Carlo WA, Garces A, Krebs NF, Hambidge KM, Saleem S, Goldenberg RL, Patel A, Hibberd PL, Esamai F, Liechty EA, Silver R, Derman RJ. A description of the methods of the aspirin supplementation for pregnancy indicated risk reduction in nulliparas (ASPIRIN) study. BMC Pregnancy Childbirth. 2017 May 3;17(1):135. doi: 10.1186/s12884-017-1312-x. PMID 28468653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, multi-country, double-masked, placebo-controlled trial of low-dose aspirin (81 mg daily) initiated between 6 weeks and 0 days of pregnancy, and 13 weeks and 6 days of pregnancy, in nulliparous women with an ultrasound confirming gestational age and a singleton viable pregnancy.
Pre-assignment Details: Participants were randomly assigned (1:1, stratified by site) to receive aspirin or placebo tablets of identical appearance, via a sequence generated centrally by the data coordinating center.
Groups:
- Intervention Arm: Daily administration of low dose (81 mg) aspirin [also known as acetylsalicylic acid (ASA], initiated between 6 0/7 weeks and 13 6/7 weeks GA and continued to 36 0/7 weeks GA.
- Placebo Arm: Identical appearing placebo beginning between 6 0/7 weeks and 13 6/7 weeks GA and continuing until 36 0/7 weeks GA or delivery.
Period: Overall Study
Arm/Group | Intervention Arm | Placebo Arm
Started | 5990 | 5986
Treated | 5943 | 5936
Included in mITT Analysis (A modified intention-to-treat (mITT) analysis was planned a priori for the primary and secondary outcomes to include only women who delivered at or after 20 weeks and were determined to be eligible after randomization. Numbers reported in the Outcomes section reflect available data and therefore do not always reflect the total population defined in the mITT.) | 5787 | 5771
Completed | 5975 | 5956
Not Completed | 15 | 30
Not completed — Lost to Follow-up | 15 | 30

BASELINE CHARACTERISTICS:
Population: Women who were eligible according to the modified intention-to-treat (mITT) criteria and included in the mITT analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Placebo Arm | Total
Number analyzed (Participants) | 5787 | 5771 | 11558
Age, Customized [Count of Participants; unit: Participants]
  Maternal Age (years): <20 years | 2233 | 2273 | 4506
  Maternal Age (years): 20-29 years | 3429 | 3372 | 6801
  Maternal Age (years): >29 years | 125 | 126 | 251
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5787 | 5771 | 11558
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Maternal Education [Count of Participants; unit: Participants]
  No formal schooling | 830 | 828 | 1658
  1-6 years of schooling | 857 | 856 | 1713
  7-12 years of scholling | 3470 | 3454 | 6924
  >= 13 years of schooling | 629 | 632 | 1261
  Missing | 1 | 1 | 2
Number of pregnancies [Count of Participants; unit: Participants]
  0 | 5274 | 5226 | 10500
  1 | 451 | 469 | 920
  2 | 62 | 76 | 138
Projected gestational age at enrollment [Median (Inter-Quartile Range); unit: weeks] | 10.1 [8.6 to 12.0] | 10.1 [8.6 to 12.0] | 10.1 [8.6 to 12.0]
Maternal Height [Mean (Standard Deviation); unit: cm] | 153.1 (6.9) | 153.1 (7.0) | 153.1 (7.0)
Maternal Weight [Mean (Standard Deviation); unit: kg] | 49.3 (8.9) | 49.2 (8.7) | 49.2 (8.8)
Maternal body-mass-index [Mean (Standard Deviation); unit: kg/m^2] | 21.0 (3.8) | 21.0 (3.6) | 21.0 (3.7)
Antenatal care visits [Median (Inter-Quartile Range); unit: visits] | 5 [4 to 6] | 5 [4 to 6] | 5 [4 to 6]
Delivery attendant [Count of Participants; unit: Participants]
  Physician | 2938 | 2908 | 5846
  Nurse or midwife | 2240 | 2239 | 4479
  Traditional birth attendant | 464 | 473 | 937
  Family, self, or other acquaintance | 142 | 147 | 289
  Missing | 3 | 4 | 7
Delivery mode [Count of Participants; unit: Participants]
  Vaginal | 4257 | 4324 | 8581
  Caesarean section | 1523 | 1440 | 2963
  Miscarriage | 0 | 0 | 0
  Medical termination of pregnancy | 5 | 4 | 9
  Missing | 2 | 3 | 5
Delivery location [Count of Participants; unit: Participants]
  Hospital | 3479 | 3494 | 6973
  Clinic or health care | 1818 | 1765 | 3583
  Home or other | 488 | 509 | 997
  Missing | 2 | 3 | 5
Site [Count of Participants; unit: Participants]
  Democratic Republic of the Congo | 655 | 665 | 1320
  Guatemala | 836 | 835 | 1671
  India (Belagavi) | 1327 | 1323 | 2650
  India (Nagpur) | 1026 | 1020 | 2046
  Kenya | 673 | 655 | 1328
  Pakistan | 771 | 762 | 1533
  Zambia | 499 | 511 | 1010

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Preterm Birth
Description: The primary outcome of this study is incidence of preterm birth, which will be defined as delivery at or after 20 0/7 weeks and prior to 37 0/7 weeks. This will be determined based on actual date of delivery in comparison to the projected estimated due date (EDD), independent of whether or not the preterm delivery is indicated or spontaneous.
Time Frame: At delivery
Population: Modified ITT; numbers reported reflect available data and therefore do not always reflect the total population defined in the mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5780 | 5764
Participants | 668 | 754
Statistical Analysis 1: Comparison: Placebo Arm; The null hypothesis is there is no treatment effect on preterm delivery; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel — A-priori threshold for statistical significance at 0.05 was specified; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.81 to 0.98]

2. Secondary Outcome: Incidence of Hypertensive Disorders of Pregnancy
Description: - Hypertensive disorders of pregnancy is defined by the characterization of evidence of a hypertensive disorder, including either preeclampsia or eclampsia occurring during the pregnancy.
Time Frame: Evidence of hypertensive disorder during the pregnancy (prior to delivery/birth)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5780 | 5764
Participants | 352 | 325
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.299, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.94 to 1.25]

3. Secondary Outcome: Incidence of Small for Gestational Age (SGA)
Description: - Small for gestational age (SGA) as defined by the INTERGROWTH-21st standard
Time Frame: At delivery or at Day 42 after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5492 | 5467
Participants | 1506 | 1564
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.171, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.90 to 1.01]

4. Secondary Outcome: Incidence of Perinatal Mortality
Description: - Incidence of Perinatal Mortality
Time Frame: At delivery or at Day 42 after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5779 | 5763
Participants | 264 | 309
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.048, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.73 to 1.00]

5. Other Pre Specified Outcome: Maternal Outcome 1 - Incidence of Vaginal Bleeding
Description: - Vaginal bleeding
Time Frame: At delivery or at Day 42 after delivery
Population: ITT population; numbers reported reflect available data and therefore do not always reflect the total population defined in the ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5933 | 5940
Participants | 214 | 246
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.125, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.73 to 1.04]

6. Other Pre Specified Outcome: Maternal Outcome 2 - Incidence of Antepartum Hemorrhage
Description: - Antepartum hemorrhage
Time Frame: At delivery or at Day 42 after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5761 | 5746
Participants | 26 | 25
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.900, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.60 to 1.79]

7. Other Pre Specified Outcome: Maternal Outcome 3 - Incidence of Postpartum Hemorrhage
Description: - Postpartum hemorrhage
Time Frame: At delivery or at Day 42 after delivery
Population: Safety population (women receiving at least one dose of drug or placebo); numbers reported reflect available data
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5928 | 5907
Participants | 54 | 43
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.274, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.25, 95% CI 2-sided [0.84 to 1.86]

8. Other Pre Specified Outcome: Maternal Outcome 4 - Incidence of Maternal Mortality
Description: - Incidence of Maternal Mortality
Time Frame: At delivery or at Day 42 after delivery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5958 | 5948
Participants | 9 | 12
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.512, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.32 to 1.78]

9. Other Pre Specified Outcome: Maternal Outcome 5 - Incidence of Late Abortion
Description: - Incidence of Late Abortion
Time Frame: At delivery or at Day 42 after delivery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5819 | 5808
Participants | 23 | 30
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.331, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.45 to 1.31]

10. Other Pre Specified Outcome: Maternal Outcome 6 - Change in Maternal Hemoglobin
Description: Hemoglobin < 7.0 gm/dl at 26-30 weeks gestation or a drop of 3.5+ gm/dl from screening to 26-30 weeks gestation
Time Frame: At enrollment, 4 weeks post enrollment, and 26-30 weeks GA.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5393 | 5398
Participants | 290 | 333

11. Other Pre Specified Outcome: Maternal Outcome 7 - Incidence of Preterm, Preeclampsia
Description: Early preterm delivery (<34 weeks) and hypertensive disorders (i.e.: preeclampsia)
Time Frame: At delivery or at Day 42 after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5780 | 5764
Participants | 8 | 21
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.38, 95% CI 2-sided [0.17 to 0.85]

12. Other Pre Specified Outcome: Fetal Outcome 1 - Incidence of Early Preterm Delivery (<34 Weeks)
Description: - Early preterm delivery (<34 weeks)
Time Frame: At delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5780 | 5764
Participants | 189 | 230
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.039, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.61 to 0.93]

13. Other Pre Specified Outcome: Fetal Outcome 2 - Incidence of Actual Birth Weight <2500g
Description: - Birth weight <2500g
Time Frame: At delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5628 | 5624
Participants | 1078 | 1153
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.073, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.87 to 1.01]

14. Other Pre Specified Outcome: Fetal Outcome 3 - Incidence of Actual Birth Weight <1500g
Description: - Birth weight <1500g
Time Frame: At delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5628 | 5624
Participants | 78 | 101
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.084, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.57 to 1.33]

15. Other Pre Specified Outcome: Fetal Outcome 4 - Incidence of Fetal Loss
Description: - Incidence of Fetal Loss
Time Frame: At delivery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5818 | 5807
Participants | 303 | 353
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.039, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.73 to 1.00]

16. Other Pre Specified Outcome: Fetal Outcome 5 - Incidence of Spontaneous Abortion
Description: - Incidence of Spontaneous Abortion
Time Frame: At delivery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5956 | 5946
Participants | 134 | 152
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.261, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.70 to 1.10]

17. Other Pre Specified Outcome: Fetal Outcome 6 - Incidence of All Stillbirth
Description: - Incidence of All stillbirth
Time Frame: At delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5780 | 5764
Participants | 141 | 166
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.141, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.68 to 1.06]

18. Other Pre Specified Outcome: Fetal Outcome 7 - Incidence of Medical Termination of Pregnancy
Description: - Incidence of Medical Termination of Pregnancy
Time Frame: At delivery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5956 | 5946
Participants | 42 | 30
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.157, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.40, 95% CI 2-sided [0.88 to 2.23]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously throughout the study (from enrollment through 6-weeks post delivery) and recorded every 2-weeks.
Description: SAEs were monitored for any event that: resulted in maternal or fetal death; was life-threatening; required hospitalization; resulted in persistent or significant disability; or any other serious or unexpected AE that the investigators felt should be reported. Specific AEs to be monitored included maternal death, upper GI bleeding, fetal anomaly, gastroschisis, post-partum hemorrhage, or antepartum hemorrhage. Other [Not Including Serious] AEs were not monitored/assessed.
Arm/Group | Intervention Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 9/5943 | 12/5936
Serious Adverse Events (participants affected / at risk) | 832/5943 | 857/5936
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=5943) | Placebo Arm (N=5936)
Maternal death (Pregnancy, puerperium and perinatal conditions) | 9 | 12
Fetal loss (Pregnancy, puerperium and perinatal conditions) | 142 | 162
Neonatal death up to 28 days (Pregnancy, puerperium and perinatal conditions) | 163 | 190
Miscarriage, abortion, or medical termination of pregnancy (Pregnancy, puerperium and perinatal conditions) | 51 | 54
Preterm labour or preterm birth evaluation before delivery (Pregnancy, puerperium and perinatal conditions) | 45 | 56
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 35 | 33
Post-partum harmorrhage (Pregnancy, puerperium and perinatal conditions) | 50 | 43
Vaginal spotting, bleeding, or leaking (Reproductive system and breast disorders) | 10 | 10
Congenital anomaly (Congenital, familial and genetic disorders) | 32 | 36
Anaemia (Blood and lymphatic system disorders) | 24 | 23
Fever or infection (Infections and infestations) | 54 | 46
Other (Pregnancy, puerperium and perinatal conditions) | 57 | 57
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 4 | 1
Pre-eclampsia or eclampsia (Pregnancy, puerperium and perinatal conditions) | 150 | 141
Hypertension admission or medical visit before delivery (Cardiac disorders) | 120 | 106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT02409680/Prot_SAP_000.pdf